CLINICAL TRIAL: NCT03663907
Title: Heart Failure Events Reduction With Remote Monitoring and eHealth Support Investigator Initiated Trial
Acronym: HERMeS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Josep Comín, Head of the Community Heart Failure Unit, Cardiology Department. MD, PhD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IDIBELL- 2017/PR190/17
Record Dates: First submitted 2018-08-28; First posted 2018-09-10 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure
Keywords: Telemedicine; Telemonitoring; Disease Management; Chronic Care Model; Transitional Care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring (Experimental): Structured follow-up in the basis of using telemedicine. Telemedicine will include daily signs and symptoms telemonitoring and structured follow-up by the means of video or audio-conference.
  Interventions: Procedure: Telemonitoring
- Usual Care (No Intervention): Patients with usual care follow-up in a heart failure program.

INTERVENTIONS:
Procedure: Telemonitoring — The system (the home tele-healthcare platform) designed jointly by engineers and clinical personal to be able daily automated selfreported symptom and weight, blood pressure and heart rate monitoring. The system allow weekly follow up through videoconferences.
  Information from the telemonitoring system is automatically downloaded to a secure Internet site for review by clinicians and nurses daily.
  Arms: Telemonitoring

SUMMARY:
The primary objective of the study is to evaluate the efficacy of a telemedicine-based follow-up strategy compared with usual care in the management of patients with chronic heart failure (HF) at high risk of clinical events.

DETAILED DESCRIPTION:
The HERMeS Trial (Heart failure Events reduction with Remote Monitoring and eHealth Support) is a multicenter, prospective, randomized, open label, observational investigator initiated study to assess the effect on cardiovascular mortality and non-fatal heart failure (HF) events of a telemedicine-based comprehensive management program for patients with chronic HF by means of remote daily telemonitoring of signs and symptoms of HF and remote structured follow-up using videoconference. The organizational characteristics of the programme and the impact in health outcomes resulting from its implementation have been previously published.

In this study we aim to compare the strategy of providing nurse-based structured follow-up to high-risk chronic HF patients through planned contacts between health care providers and patients and/or caregivers in the basis of face-to-face on-site encounters (usual care) or provide the planned care using telemedicine with the combination of remote daily monitoring of signs and symptoms of HF (telemonitoring) and delivery of structured nurse-based follow-up health care using videoconference (tele-intervention).

The main hypothesis of the study is that daily telemonitoring of clinical variables and symptoms in high-risk patients with HF allows early detection of decompensations by decreasing the number of fatal cardiovascular events or non-fatal HF events. As a secondary hypothesis we assume that tele-intervention using telemedicine may help to optimise neurohormonal treatment and deliver appropriate education to high-risk patients with HF; and delivery of care in high risk patients with HF through the combination of remote monitoring and tele-intervention may translate into a reduction of fatal and non fatal HF-related events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Patients discharged from a heart failure hospitalization within 30 days of enrollment into the study or in the process of discharge planning.
* Heart Failure diagnosis according to European Society of Cardiology (ESC) criteria.
* Written informed consent must be obtained before any assessment is performed.
* Patients receiving oral standard medication for chronic heart failure (CHF).
* All patients will be eligible regardless the level of left ventricular ejection fraction (LVEF).

Exclusion Criteria:

* Age<18 years old.
* Participation in another clinical trial.
* Moderate or severe cognitive impairment without a competent caregiver.
* Lack of social support.
* Institutionalized patients.
* Life expectancy less than 1 year (excluding HF).
* Candidates for home-based or institutional end-of-life care.
* Serious psychiatric illness.
* Planned cardiac surgery.
* Planned Heart transplantation or left ventricular assist device (LVAD) implant.
* Patients in hemodialysis program.
* Death before hospital discharge.
* The patient is unable or unwilling to give the informed consent to participate.
* The patient is considered not to be an adequate candidate for this study according to the decision of the local investigator.
* Unstable patients with signs of fluid overload or low cardiac output.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Occurrence of cardiovascular death or non-fatal heart failure events. | Six months after inclusion of the patient
  Occurrence of cardiovascular death or non-fatal heart failure events (time to first event) during a follow-up period of 6 months. Non-fatal heart failure event is defined as a new episode of worsening of symptoms and signs consistent with acute decompensated HF requiring intravenous decongestive therapy (e.g. diuretics) either on an outpatient basis (day-case HF hospital) or in the emergency department (<24 hours) or requiring unplanned hospital admission (>24 hours) or complicating the course of a non-cardiovascular admission.

SECONDARY OUTCOMES:
Readmission (all-cause, HF and cardiovascular) rate and total number. | Six months after inclusion of the patient.
  Comparison of both strategies at the end of follow-up.
Days in hospital (all-cause, HF and cardiovascular). | Six months after inclusion of the patient.
  Comparison of both strategies at the end of follow-up.
Rate of emergency visits. | Six months after inclusion of the patient.
  Comparison of both strategies at the end of follow-up.
Rate of non-fatal HF events. | Six months after inclusion of the patient.
  Comparison of both strategies at the end of follow-up.
Mortality for any cause and cardiovascular mortality. | Six months after inclusion of the patient.
  Comparison of both strategies at the end of follow-up.
Improvement of self-care using a validated scale (European Heart Failure Self-Care Behavior Scale). | Six months after inclusion of the patient.
  Comparison of both strategies at the end of follow-up.
Improvement of quality of life using a validated questionnaire (EUROQOL - 5D). | Six months after inclusion of the patient.
  Comparison of both strategies at the end of follow-up.
Patient satisfaction using a Likert-type scale. | Six months after inclusion of the patient.
  Comparison of both strategies at the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Comín Colet, MD,PhD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- University Hospital Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Yun S, Comin-Colet J, Calero-Molina E, Hidalgo E, Jose-Bazan N, Cobo Marcos M, Soria T, Llacer P, Fernandez C, Garcia-Pinilla JM, Cruzado C, Gonzalez-Franco A, Garcia-Marina EM, Morales-Rull JL, Sole C, Garcia-Romero E, Nunez J, Civera J, Fernandez C, Faraudo M, Moliner P, Formiga F, de-Juan Baguda J, Zegri-Reiriz I, Verdu-Rotellar JM, Vela E, Monterde D, Piera-Jimenez J, Carot-Sans G, Enjuanes C; HERMeS trial investigators group. Evaluation of mobile health technology combining telemonitoring and teleintervention versus usual care in vulnerable-phase heart failure management (HERMeS): a multicentre, randomised controlled trial. Lancet Digit Health. 2025 May;7(5):100866. doi: 10.1016/j.landig.2025.02.006. Epub 2025 May 14. PMID 40374486